CLINICAL TRIAL: NCT01540760
Title: A Phase Ib, Single-Center, Randomized, Placebo-Controlled, Double-Blind Multiple Ascending-Dose Study to Investigate the Safety, Pharmacokinetics, and Immunogenicity of Subcutaneous MCAF5352A in Healthy Volunteers
Brief Title: A Study of MCAF5352A in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GA28006
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MCAF5352A (Experimental)
  Interventions: Drug: MCAF5352A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MCAF5352A — Multiple ascending doses
  Arms: MCAF5352A
Drug: Placebo — Matching MCAF5352A, multiple doses
  Arms: Placebo

SUMMARY:
This single-center, randomized, placebo-controlled, double-blind, multiple ascending dose study will evaluate the safety, pharmacokinetics and immunogenicity of MCAF5352A in healthy volunteers. Subjects will be randomized to receive either MCAF5352A or placebo on Days 1, 15 and 29.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, 18 - 55 years of age
* Subjects in good health as determined by screening medical history, physical examination, vital signs, 12-lead ECG and laboratory tests
* Body weight between 45 kg and 110 kg
* Female subjects must be willing to use two effective methods of contraception from screening to a minimum of 4 months after the last dose of study drug

Exclusion Criteria:

* Pregnant or lactating women
* Positive for hepatitis B, hepatitis C or HIV infection
* History of significant chronic or recurrent infections
* History of clinically significant drug allergy and/or a known hypersensitivity to protein therapeutics or formulation components or a related drug
* History of alcohol or drug abuse within 12 months prior to Day 1, or evidence of such abuse
* Subjects who have previously received the study drug
* Participation in a clinical trial within 4 weeks prior to Day 1 or use of any experimental or biologic therapy within 12 weeks prior to Day 1 or within 5 half-lives of the product, whichever is greater

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 5 months

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve | Pre-dose and 5 time points up to 14 days post-dose
Immunogenicity: Serum MCAF5252A antibodies | Days 1, 29, 50, 78, 106 and 134

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Québec, Quebec, Canada